CLINICAL TRIAL: NCT05763160
Title: An Open Label Phase 2 Study to Evaluate the Safety and Efficacy of a Second Treatment Session of RZL-012 Into Submental Fat in Subjects Seeking Further Improvement
Brief Title: An Open-label Study That Will Test a Second Treatment Session of RZL-012.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZL-012-SMF-2nd-P2US-001
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-02

CONDITIONS: Submental Fat
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Intervention Model Description: Second injection session of RZL-012 will be administered to subjects who previously treated with RZL-012 in submental fat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RZL-012 50mg/ml (Experimental)
  Interventions: Drug: RZL-012

INTERVENTIONS:
Drug: RZL-012 — Ready to use drug product for injection into the subcutaneous fat

SUMMARY:
This is a Phase 2, open-label study in which subjects seeking further improvement of their SMF will be treated with a second treatment session of RZL-012.

The second treatment session will be offered to subjects previously treated with RZL-012 under protocols RZL-012-SMF-SWMTG-P2US-001 or RZL-012-SMFC-P2US-001. Subjects who fully completed either of the trials and whose C-CAT score is 2, 3 or 4 will be eligible to participate in the new trial.

For each subject, the study will consist of a screening period, baseline period in which subjects will receive a second treatment session of RZL-012 and a follow-up period. RZL-012 will be administered during a single treatment session via multiple injections into the submental area under the chin. Subjects will thereafter be monitored for safety and efficacy for at least 84 days.

DETAILED DESCRIPTION:
Screening Period:

Subjects will be eligible to undergo screening after successful completion of (defined as completion of the day 84 visit) of either RZL-012-SMF-SWMTG-P2US-001 or RZL-012-SMFC-P2US-001 studies. Subjects will undergo screening within 28 days prior 2nd RZL session. During the screening period, subjects will be assessed for study eligibility by evaluation of subjects' SMF using S-CAT, C-CAT, SIQ8, biochemistry blood tests, 2D photography.

Day 0/Baseline:

Subjects will receive a second multi-injection treatment of RZL-012 on Day 0. AEs will be recorded. Subjects will be asked about their pain levels using VAS.

Day 1-Day 84 Follow-Up Period Subjects will return to the site for study visits on Days 1, 7, 28, 56 and 84 for efficacy and safety assessments.

Safety assessments will include vital signs, labs, AEs severity assessment, and treatment area evaluation. Treatment area evaluations will include evaluation of edema, bruising, dysphasia, dysphonia, erythema, dyspigmentation, induration, numbness, pain, paresthesia, pruritus, skin ulceration and necrosis, injury to the marginal mandibular nerve, vascular and nerve injury, and tissue damage to nearby vulnerable anatomic structures. Swelling severity will be assessed as a function of time. Pain will be assessed using the VAS. Concomitant medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible for this study, he or she must meet all of the following criteria:

1. Is a male or female subject between the ages of 18 and 65 years, inclusive.
2. Previously treated with RZL-012 under protocols RZL-012-SMF-SWMTG-P2US-001 or RZL-012-SMFC-P2US-001 and whose current C-CAT score is 2, 3 or 4
3. Who successfully completed (as in completed the day 84 visit) the RZL-012-SMF-SWMTG-P2US-001 or RZL-012-SMFC-P2US-001 studies.
4. Has body mass index (BMI) between >22 kg/m2 and <40 kg/m2.
5. Has SMF bulge that is contiguous and can receive between 16 to 36 injections distanced 1 centimeter (cm) from each other according to the injection grid.
6. Has stable weight, with no fluctuation of >5 kg in the past 12 months.
7. If female, is not pregnant or breastfeeding based on the following:

   1. agree to the use of highly effective contraceptive methods for at least 2 weeks before baseline until 4 weeks after the last day of study drug and a negative serum pregnancy test (ß-hCG) at screening and negative urine pregnancy test at baseline; or
   2. is abstaining
   3. is of nonchildbearing potential defined as clinically infertile as the result of surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy); or
   4. is confirmed postmenopausal status (defined as either having amenorrhea for ≥ 12 consecutive months without another cause or documented serum follicle-stimulating hormone (FSH) level > 40 mIU/mL or another documented medical condition (e.g., was born without a uterus)) NOTE: The following are considered highly effective contraceptive methods: hormonal oral contraceptives, injectables, and patches; intrauterine devices; double-barrier methods (synthetic condom, diaphragm, or cervical cap used with spermicidal foam, cream, or gel); and male partner sterilization.
8. If male (with or without vasectomy), agree to the use of highly effective contraceptive methods as listed above in criteria 7 as well as to use a barrier method, e.g. condom, from study check-in until 7 days after drug injection.
9. Is willing to avoid strenuous exercise for seven (7) days post treatment.
10. Can adhere to the visit schedule and protocol requirements and be available to complete the study.
11. Is willing and able to sign an Institutional Review Board (IRB) approved informed consent form (ICF) indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

* Subjects must NOT meet any of the following Exclusion criteria to be eligible for enrollment:

  1. Is unable to tolerate subcutaneous injections.
  2. Any subject who had any treatment related SAE's or allergic reactions to treatment in the previous RZL-012 studies.
  3. Has any systemic disease including but not limited to gastritis or ulcers, renal dysfunction, hypertension, liver disease, glaucoma, diabetes and/or cardiovascular disease, regardless of whether the condition is controlled with medication.
  4. Has skin laxity (i.e., elastosis, skin crepiness, skin redundancy, skin draping, vertical and/or horizontal skin bands and folds, blunting of cervical mental angle, loss of opposition of skin to underlying neck structures due to skin laxity) that could obscure the evaluation and treatment of SMF.
  5. Has any scars, unshaven hair, tattoos, facial hair, or jewelry on or near the proposed treatment area.
  6. Has presence of structures or confounding factors that may interfere with assessing SMF such as but not limited to enlarged submandibular salivary and/or parotid glands, micrognathia, chin implant, soft tissue volume augmentation of chin and/or jawline, pronounced platysmal bands and deep necklace lines or presence of facial jowls that could obscure the evaluation of SMF.
  7. Has a fat bulge under the chin that is too large to be adequately treated by 36 contiguous injections on a 1cm grid .
  8. Has a fat bulge under the chin that is of an insufficient volume to allow 16 injections within a contiguous 1 cm grid.
  9. Has significant history or current evidence of a medical, psychological, or other disorder that, in the Investigator's opinion, would preclude enrollment in the study.
  10. Has an active bacterial, fungal, or viral infection in the proposed treatment area.
  11. Has a pre-existing skin condition in the submental region that, at the Investigator's discretion, may confound evaluation or analysis.
  12. Has previously had treatments or surgery in the submentum, such as but not limited to, focused ultrasound, radiofrequency, cryolipolysis, liposuction, sodium deoxycholate, or neck lift.
  13. Has pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia, or facial nerve palsy.
  14. Has Dercum's Disease.
  15. Has allergic reactions to injectables
  16. Has any pre-existing medical condition other than increased SMF that, at the Investigator's discretion, may result in increased submental fullness, such as but not limited to, thyroid enlargement, goiter, cervical lymphadenopathy, etc.
  17. Has a planned fat reduction procedure of any variety to the submental region for the duration of the study.
  18. Has medication or a history of coagulopathy.
  19. Has a history or family history of venous thrombotic disease.
  20. Has been treated chronically at least three (3) months prior to study entry with systemic steroids or immunosuppressive drugs.
  21. Has been treated chronically at least one (1) week prior to study entry with non-steroidal anti-inflammatory drugs (NSAIDs)
  22. Has used anticoagulation therapies that may increase bleeding or bruising (i.e., aspirin, ibuprofen/Celecoxib, warfarin, vitamins, and herbal preparations) for seven (7) days prior to treatment.
  23. Has had treatment with botulinum toxin injections in the neck or chin area within nine (9) months prior to screening.
  24. Current participation or participation within three (3) months prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse events follow up | 84 days
  Safety assessments will include vital signs, labs, AEs severity assessment, and treatment area evaluation. Treatment area evaluations will include evaluation of edema, bruising, dysphasia, dysphonia, erythema, dyspigmentation, induration, numbness, pain, paresthesia, pruritus, skin ulceration and necrosis, injury to the marginal mandibular nerve, vascular and nerve injury, and tissue damage to nearby vulnerable anatomic structures. Swelling severity will be assessed as a function of time. Pain will be assessed using the VAS. Concomitant medications will be recorded

SECONDARY OUTCOMES:
Efficacy -Change in score according to Clinician chin assessment tool (C-CAT) | 84 days
  • Proportion of subjects who have at least a 1-grade improvement in C-CAT on Day 84 versus baseline in subjects receiving a second treatment session of RZL-012. Baseline is defined as the C-CAT assessment made immediately prior to the second treatment session

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No